CLINICAL TRIAL: NCT02314559
Title: A Psychomotor Recuperation Study After Deep Sedation for Colonoscopy Between Target Controlled and Manual Titration of Propofol.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head of anesthesiology department, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CHUB Mental Recup 001
Record Dates: First submitted 2014-12-05; First posted 2014-12-11 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Colonoscopy (Ambulatory Patients)
Keywords: propofol; colonoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (manual titration) (Experimental)
  Interventions: Drug: Manual titration of propofol
- Propofol (target controlled infusion) (Active Comparator)
  Interventions: Drug: Target controlled infusion of propofol

INTERVENTIONS:
Drug: Manual titration of propofol — One group will be sedated with a manual titration technique: here the titration of propofol is done manually by the anesthetist. Dosages may range between 50 and 400mg, given by boluses of 20-50mg.
  Arms: Propofol (manual titration)
Drug: Target controlled infusion of propofol — The other group will be sedated with a target controlled infusion technique (pump, marsh or Schneider). The anesthetist can titrate indirectly by adjusting the target controlled infusion to achieve adequate sedation. The concentrations of propofol may vary between 2 and 6 µg/ml, achieved by increments of 0.5-1.5 µg/ml.
  Arms: Propofol (target controlled infusion)

SUMMARY:
Deep sedation with propofol for ambulatory colonoscopy has become standard clinical practice.To achieve the necessary (e.g.: no excessive movement and no awareness) level of sedation during colonoscopy, propofol can be titrated by hand, continuous infusion or by target controlled infusion.

The aim of the investigators is to evaluate sedation efficacy and recovery between two groups of ambulatory patients having a colonoscopy: one group will receive a manual titration of propofol, the other group a target controlled infusion (TCI) of propofol. The investigators will evaluate both groups before, during and after colonoscopy for adverse events, quality of sedation and recovery. When patients are estimated to be ready for discharge, they will also be subjected to a cognitive and a psychomotoricity test.

DETAILED DESCRIPTION:
Deep sedation with propofol for ambulatory colonoscopy has become standard clinical practice. Fewer adverse events and a faster wake up time than with the use of benzodiazepines are proven. A growing group of patients are subjected to this examination for diagnostic and screening purposes.

In most cases, patients can return home after a short recovery time, under the supervision of an accompanying person. Often, no residual effects are clinically detectable. Some studies advocate that driving skills recover quickly. Current guidelines however, insist to avoid driving or using public transportation alone for at least 12 hours (24 hours if other sedatives are used).

To achieve the necessary (e.g.: no excessive movement and no awareness) level of sedation during colonoscopy, propofol can be titrated by hand, continuous infusion or by target controlled infusion. Only one study, to the investigators knowledge, compares efficacy between manual titration and target controlled infusion of propofol in combination with fentanyl for bidirectional endoscopy.

The aim of the investigators is to evaluate sedation efficacy and recovery between two groups of ambulatory patients having a colonoscopy: one group will receive a manual titration of propofol, the other group a target controlled infusion (TCI) of propofol. The investigators will evaluate both groups before, during and after colonoscopy for adverse events, quality of sedation and recovery. When patients are estimated to be ready for discharge, they will also be subjected to a cognitive and a psychomotoricity test.

To evaluate cognitive function, the investigators will use the digit symbol substitution test. The digit symbol substitution test is popular for detecting deterioration in concentration. Here for 90 seconds, a test subject is asked to change a number in a symbol.

As psychomotor test, the investigators chose a choice reaction time test for its sensitivity to detect minor changes after propofol sedation. This test has also validity in alcohol intoxication. A simple reaction time test is also included for its easy applicability and obtainability in everyday practive. Test results will be compared to see if there is a correlation with the choice reaction time tests.

ELIGIBILITY:
Inclusion Criteria:

* All patients subjected to deep sedation in ambulant care, having a colonoscopy
* ASA 1-3

Exclusion Criteria:

* Dementia.
* Gastroscopy planned at the same time.
* Allergies to propofol
* All cases were a 'full stomach' is suspected (gastric banding)
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2015-02; Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Digit Symbol Substitution test score | 24 hours
  The digit symbol substitution test score wil be compared between the propofol manual titration and the propofol target controled infusion groups. This test will evaluate cognitive function.
PADS score | 24 hours
  Time and fitness to discharge will be evaluated with the PADS score. This will be done at discharge of the patient, after the colonoscopy.
Choice reaction time test score | 24 hours
  The choice reaction time test score will be compared between the propofol manual titration and the propofol target controlled infusion groups. The groups will be tested before the colonoscopy and every 10 minutes after waking up, up to the discharge of the patient. This test is used to evaluate the psychomotoricity of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Schmartz, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riphaus A, Geist F, Wehrmann T. Endoscopic sedation and monitoring practice in Germany: re-evaluation from the first nationwide survey 3 years after the implementation of an evidence and consent based national guideline. Z Gastroenterol. 2013 Sep;51(9):1082-8. doi: 10.1055/s-0033-1335104. Epub 2013 Sep 10. PMID 24022202
- [Background] Cohen LB, Wecsler JS, Gaetano JN, Benson AA, Miller KM, Durkalski V, Aisenberg J. Endoscopic sedation in the United States: results from a nationwide survey. Am J Gastroenterol. 2006 May;101(5):967-74. doi: 10.1111/j.1572-0241.2006.00500.x. PMID 16573781
- [Background] Carlsson U, Grattidge P. Sedation for upper gastrointestinal endoscopy: a comparative study of propofol and midazolam. Endoscopy. 1995 Mar;27(3):240-3. doi: 10.1055/s-2007-1005678. PMID 7664702
- [Background] Qadeer MA, Vargo JJ, Khandwala F, Lopez R, Zuccaro G. Propofol versus traditional sedative agents for gastrointestinal endoscopy: a meta-analysis. Clin Gastroenterol Hepatol. 2005 Nov;3(11):1049-56. doi: 10.1016/s1542-3565(05)00742-1. PMID 16271333
- [Background] Riphaus A, Gstettenbauer T, Frenz MB, Wehrmann T. Quality of psychomotor recovery after propofol sedation for routine endoscopy: a randomized and controlled study. Endoscopy. 2006 Jul;38(7):677-83. doi: 10.1055/s-2006-925244. PMID 16810592
- [Background] Horiuchi A, Nakayama Y, Katsuyama Y, Ohmori S, Ichise Y, Tanaka N. Safety and driving ability following low-dose propofol sedation. Digestion. 2008;78(4):190-4. doi: 10.1159/000187118. Epub 2008 Dec 18. PMID 19092246
- [Background] Dumonceau JM, Riphaus A, Aparicio JR, Beilenhoff U, Knape JT, Ortmann M, Paspatis G, Ponsioen CY, Racz I, Schreiber F, Vilmann P, Wehrmann T, Wientjes C, Walder B; NAAP Task Force Members. European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates, and the European Society of Anaesthesiology Guideline: Non-anesthesiologist administration of propofol for GI endoscopy. Endoscopy. 2010 Nov;42(11):960-74. doi: 10.1055/s-0030-1255728. Epub 2010 Nov 11. PMID 21072716
- [Background] Chiang MH, Wu SC, You CH, Wu KL, Chiu YC, Ma CW, Kao CW, Lin KC, Chen KH, Wang PC, Chou AK. Target-controlled infusion vs. manually controlled infusion of propofol with alfentanil for bidirectional endoscopy: a randomized controlled trial. Endoscopy. 2013 Nov;45(11):907-14. doi: 10.1055/s-0033-1344645. Epub 2013 Oct 28. PMID 24165817
- [Background] Grant SA, Murdoch J, Millar K, Kenny GN. Blood propofol concentration and psychomotor effects on driving skills. Br J Anaesth. 2000 Sep;85(3):396-400. doi: 10.1093/bja/85.3.396. PMID 11103180
- [Background] Grant SA, Millar K, Kenny GN. Blood alcohol concentration and psychomotor effects. Br J Anaesth. 2000 Sep;85(3):401-6. doi: 10.1093/bja/85.3.401. PMID 11103181
- [Background] Trevisani L, Cifala V, Gilli G, Matarese V, Zelante A, Sartori S. Post-Anaesthetic Discharge Scoring System to assess patient recovery and discharge after colonoscopy. World J Gastrointest Endosc. 2013 Oct 16;5(10):502-7. doi: 10.4253/wjge.v5.i10.502. PMID 24147194
- [Background] Deary IJ, Liewald D, Nissan J. A free, easy-to-use, computer-based simple and four-choice reaction time programme: the Deary-Liewald reaction time task. Behav Res Methods. 2011 Mar;43(1):258-68. doi: 10.3758/s13428-010-0024-1. PMID 21287123